CLINICAL TRIAL: NCT06145295
Title: Understanding the Effectiveness of an Online Support Group in Enhancing Recovery Identity and Health-Related Quality of Life of Middle-aged and Older Ovarian Cancer Patients: A Randomized Controlled Trial
Brief Title: The Effectiveness of an Online Support Group in Enhancing Recovery Identity and Health-Related Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Jianan Zhao, Principal Investigator, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 507079
Record Dates: First submitted 2023-11-15; First posted 2023-11-24 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experiment group (online support group) (Experimental): The experimental group engaged with the mobile application use for four weeks, with specific tasks including completing the four mandatory courses within one month and submitting at least two health records and online posts every week.
  Interventions: Behavioral: mobile online support group (experiment group)
- control group (Other): The control group participates in the offline group intervention that last for four weeks. Participants in the control group will participant in four weekly workshop that last between 1 hour to 1.5 hours.
  Interventions: Behavioral: offline support group (control group)

INTERVENTIONS:
Behavioral: mobile online support group (experiment group) — The experimental group engaged with the mobile application use for four weeks, with specific tasks including completing the four mandatory courses within one month and submitting at least two health records and online posts every week.
  Arms: experiment group (online support group)
Behavioral: offline support group (control group) — The control group participates in the offline group intervention that last for four weeks. Participants in the control group will participant in four weekly workshop that last between 1 hour to 1.5 hours.
  Arms: control group

SUMMARY:
Background Ovarian cancer poses challenges for middle-aged and older patients, impacting physical and self-conceptual aspects. A research gap exists on the impact of online support groups (SPs) on identity synthesis and Health-Related Quality of Life (HRQOL) for these patients.

Objective To assess the feasibility and efficacy of an online SG in influencing recovery identity and HRQOL in middle-aged and older ovarian cancer patients (MDOCP).

Method A four-week randomized controlled trial, followed by a three-month evaluation, was conducted, employing a mobile online SG and an offline SG both grounded in The Social Identity Model of Identity Change. Recovery identity, HRQOL, and participant engagement were utilized to evaluate the feasibility and efficacy of interventions.

ELIGIBILITY:
Inclusion Criteria:

* Older than 44 years old
* diagnosis of ovarian cancer
* expected survival time of greater than four months
* fluent in using smartphones and the WeChat mini program
* normal cognitive function
* capability to participate in follow-up surveys.

Exclusion Criteria:

* were currently participating in or had previously participated in other mental treatment groups
* had been diagnosed with any other type of cancer.

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-10-25 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Illness identity | Data collection occurred at three time points: before the intervention, immediately after the intervention, and at a three-month follow-up
  The acceptance of illness identity was measured using the Illness Identity Questionnaire's acceptance sub-scale, consisting of 6 items (Oris et al., 2016).
Maintenance of identity | Data collection occurred at three time points: before the intervention, immediately after the intervention, and at a three-month follow-up
  The maintenance of former social identities was measured using the Maintenance of Group Memberships sub-scale of Exeter Identity Transition Scales (Haslam et al., 2008), encompassing 4 items.
New identity | Data collection occurred at three time points: before the intervention, immediately after the intervention, and at a three-month follow-up
  The new meaningful social identity was measured using the New Group Memberships sub-scale of the Exeter Identity Transition Scales, which includes 4 questions. Responses were rated on a scale from 1 to 5, with higher scores indicating a higher level of acceptance of the identity.

SECONDARY OUTCOMES:
Health related quality of life | Data collection occurred at three time points: before the intervention, immediately after the intervention, and at a three-month follow-up
  Health related quality of life was measured using the Short Form Health Survey 12 (SF-12) (Jakobusson, 2007), which includes twelve questions. Each item is transformed into a scale ranging from 0 to 100 according to a specific scoring algorithm. These scores are then aggregated to generate two summary scores: the Physical Component Summary (PCS) and the Mental Component Summary (MCS). The resulting scores are norm-based, comparing an individual's health status to population norms. Health related quality of life is calculate as the summary of PCS and MCS. Higher scores indicate better health related quality of life, with scores around 50 representing the average.

CONTACTS AND LOCATIONS:
Overall Officials: Ting Han, Ph.D., Study Chair — Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai Jiao Tong Universiy, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon reasonable request to the researcher (the private information of the participant will be removed).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After the article is accepted
Access Criteria: The data will be available upon reasonable request to the researcher (the private information of the participant will be removed).

REFERENCES:
- [Derived] Zhao J, Zhu D, Yang Y, Tian C, Liu C, Chang F, Han T. Understanding the effectiveness of an online support group in enhancing recovery identity and health-related quality of life of middle-aged and older ovarian cancer patients: A randomized controlled trial. Psychol Trauma. 2025 Jun;17(Suppl 1):S196-S205. doi: 10.1037/tra0001929. PMID 40569778

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-16): https://cdn.clinicaltrials.gov/large-docs/95/NCT06145295/Prot_SAP_000.pdf